CLINICAL TRIAL: NCT02129933
Title: A Pilot Intervention Study for the Use of VEGF-targeted Fluorescence Near-Infrared (NIR) Endoscopy in (Pre)Malignant Esophageal Lesions
Brief Title: VEGF-targeted Fluorescence Near-Infrared (NIR) Endoscopy in (Pre)Malignant Esophageal Lesions
Acronym: VICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL45554.042.14; 2013-003003-19 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-05-02 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer; Dysplasia
Keywords: EAC; HGD; Esophagus
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tracer bevacizumab-IRDye800CW (Experimental): Two days prior to the fluorescence endoscopy procedure (with the near infrared fluorescence endoscopy platform), all patients will receive the fluorescent tracer bevacizumab-IRDye800CW intravenously.
  *amendement June 2015: topical administration of bevacizumab-800CW
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Near infrared fluorescence endoscopy platform

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Intravenous administration of a microdose (4.5mg, subtherapeutic) of Bevacizumab-IRDye800CW 2 days prior to the fluorescence endoscopy procedure.
  * amendment June 2015: topical administration bevacizumab-800CW (100ug/ml)
  Other Names: Beva-800CW; Bevacizumab-800CW; Avastin-800CW (Roche)
Device: Near infrared fluorescence endoscopy platform — A flexible fiber-bundle is attached with its proximal end to a camera which can detect near infrared fluorescent light. The distal end is inserted into the working channel of a clinical video endoscope to visualize the luminal wall. The fluorescent imaging will be performed prior and post the endoscopic resection (within the same endoscopic session)

SUMMARY:
To improve detection of esophageal (pre)malignant lesions during surveillance endoscopy of patients at risk of developing malignancies, for example in Barrett's Esophagus (BE), there is a need for better endoscopic visualization and the ability for targeted biopsies. Optical molecular imaging of neoplasia associated biomarkers could form a promising technique to accommodate this need. It is known that the biomarker Vascular Endothelial Growth Factor (VEGF) is overexpressed in dysplastic and neoplastic areas in BE segments versus normal tissue and has proven to be a valid target for molecular imaging. The University Medical Center Groningen (UMCG) developed a fluorescent tracer by labeling the VEGF-targeting humanized monoclonal antibody bevacizumab, currently used in anti-cancer therapy, with the fluorescent dye IRDye800CW. We hypothesize that when bevacizumab-IRDye800CW is administered, it accumulates in VEGF expressing high grade dysplasia (HGD) and esophageal adenocarcinoma (EAC), enabling early cancer visualization using a newly developed fluorescent NIR fiber-bundle. This hypothesis will be tested in this pilot intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Identified HGD or intramucosal EAC (T1) and therefore candidate for endoscopic mucosal resection therapy
* Mentally competent person, 18 years or older.
* Written informed consent.
* Adequate potential for follow-up.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Submucosal and invasive EAC; EAC with tumor-classification other than T1.
* Concurrent (uncontrolled) medical conditions which disqualify for an endoscopic mucosal resection procedure.
* Previously performed therapeutic endoscopic procedures.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
NIR fluorescent signal in vivo (prior to EMR) | 1 day (endoscopy-day)
  Evaluating presence of specific fluorescent signal in (pre)malignant esophageal lesion in vivo, with use of Near Infrared (NIR) fluorescence endoscopy platform.

SECONDARY OUTCOMES:
Number of participants with adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR). | Two days prior and up to 1 week after administration of tracer
  Data collection as a measure of safety and tolerability regarding administration of Bevacizumab-IRDye800CW
VEGF expression ex vivo | up to 1 year
  Correlation between specific fluorescent signal in vivo and ex vivo (observed with near-infrared fluorescence endoscopy) and VEGF expression ex vivo (immunohistochemistry).
NIR fluorescent signal in vivo (wound bed, post EMR) | 1 day (endoscopy-day)
  Presence of specific fluorescence signal in correlation to histological evaluation of specimen (resection margins)
NIR fluorescent signal ex vivo (biopsy and EMR specimen) | up to 1 year
  Evaluation of specific fluorescent signal ex vivo in correlation with observed fluorescence signal during endoscopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter B Nagengast, PharmD MD PhD, Principal Investigator — University Medical Center Groningen; Frans TM Peters, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Nagengast WB, Hartmans E, Garcia-Allende PB, Peters FTM, Linssen MD, Koch M, Koller M, Tjalma JJJ, Karrenbeld A, Jorritsma-Smit A, Kleibeuker JH, van Dam GM, Ntziachristos V. Near-infrared fluorescence molecular endoscopy detects dysplastic oesophageal lesions using topical and systemic tracer of vascular endothelial growth factor A. Gut. 2019 Jan;68(1):7-10. doi: 10.1136/gutjnl-2017-314953. Epub 2017 Dec 15. No abstract available. PMID 29247063